CLINICAL TRIAL: NCT04038788
Title: The Effects of High-Definition High-Frequency Transcranial Random Noise Stimulation Over Bilateral Prefrontal Cortex on Illness Symptoms, Clinical Outcomes, Autonomic Function and Brain Oscillatory Activity in Schizophrenia Patients
Brief Title: Add-on HD Hf-tRNS Over Bilateral DLPFC for Treating Patients With Schizophrenia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tri-Service General Hospital (Other)
Responsible Party: Principal Investigator, Hsin-An Chang, MD, Attending Psychiatrist, Department of Psychiatry, Principal Investigator, Associate Professor, Tri-Service General Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2-107-03-001
Record Dates: First submitted 2019-07-18; First posted 2019-07-31 (Actual); Last update posted 2019-07-31 (Actual); Status verified 2019-07

CONDITIONS: Schizophrenia; Schizoaffective Disorder; Psychotic Symptoms; Neurocognitive Dysfunction; Insight Impaired; Quality of Life; Psychosocial Impairment; Autonomic Imbalance; EEG With Abnormally Slow Frequencies
MeSH Terms: conditions — Schizophrenia; Psychotic Disorders; Cognition Disorders

STUDY DESIGN:
Intervention Model Description: In active tRNS condition, random noise was delivered by a battery-operated device (Eldith DC stimulator Plus, neuroConn, Ilmenau, Germany) via 5 carbon rubber electrodes (1 cm radius, high-definition 4 × 1 rings configuration with a gel layer of 2.0 mm), with 2 mA amplitude, offset at 1 mA, frequency 100-640 Hz, for 20 min with 15 s ramp-in/ramp-out. The combined impedance of all electrodes was kept below 15 kΩ, as measured by NeuroConn DC stimulator Plus device, using electrolyte gel. The anode was placed over International 10-10 electrode position AF3 (a point midway between F3 and Fp1), with cathodes (reference electrodes) at AF4, F2, F6 and FC4. Stimulation was applied at an intensity of 2 milliampere (mA) for 20 min, twice-daily on 5 consecutive weekdays.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: In sham stimulation, the current was turned on for 30 sec and then ramped down to 0 mA.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Active tRNS (Active Comparator): In active tRNS condition, random noise was delivered by a battery-operated device (Eldith DC stimulator Plus, neuroConn, Ilmenau, Germany) via 5 carbon rubber electrodes (1 cm radius, high-definition 4 × 1 rings configuration with a gel layer of 2.0 mm), with 2 mA amplitude, offset at 1 mA, frequency 100-640 Hz, for 20 min with 15 s ramp-in/ramp-out. The combined impedance of all electrodes was kept below 15 kΩ, as measured by NeuroConn DC stimulator Plus device, using electrolyte gel. The anode was placed over International 10-10 electrode position AF3 (a point midway between F3 and Fp1), with cathodes (reference electrodes) at AF4, F2, F6 and FC4. Stimulation was applied at an intensity of 2 milliampere (mA) for 20 min, twice-daily on 5 consecutive weekdays. All patients in the active stimulation group were maintained on their antipsychotic medications throughout the study period.
  Interventions: Device: HD hf-tRNS
- Sham treatment (Sham Comparator): In sham stimulation, the current was turned on for 30 sec and then ramped down to 0 mA. All patients in the sham group were maintained on their antipsychotic medications throughout the study period.
  Interventions: Device: HD hf-tRNS

INTERVENTIONS:
Device: HD hf-tRNS — See detail in arm/group descriptions regarding the intervention.

SUMMARY:
The study aimed to investigate the effects of high-definition transcranial random noise stimulation over bilateral prefrontal cortex on psychopathological symptoms, other clinical outcomes, autonomic functioning ,and brain oscillatory activity in schizophrenia patients.

DETAILED DESCRIPTION:
Negative symptoms of schizophrenia include blunted affect, avolition-apathy, alogia and anhedonia-asociality and are closely linked to neurocognitive deficits. Negative symptoms and neurocognitive impairments are associated with poor functional outcomes. Prefrontal cortical dysfunction, particularly hypoactivity of the dorsolateral prefrontal cortex (DLPFC) has consistently been reported in schizophrenia and suggested to underlie the pathophysiology of negative symptom and neurocognitive impairment. Atypical antipsychotics, the mainstream treatment for schizophrenia, are known to show little effect on patients' hypofrontality and some of them (e.g., strong dopamine receptor antagonists and clozapine) are even associated with a decrease in prefrontal activation. Furthermore, good evidence that atypical antipsychotics have any beneficial effect on negative symptoms or neurocognitive impairments is still lacking. Currently, negative symptoms and cognitive deficits remain the most important unmet therapeutic needs in schizophrenia, which have driven the development of novel and effective treatments targeting the core pathophysiological features of the deficits, e.g., non-invasive brain stimulation (NIBS) of DLPFC.

Transcranial random noise stimulation (tRNS) is a neuromodulation technique that applies a weak alternating current over the brain cortex at random frequencies (0.1- 640 Hz), i.e., the current oscillating randomly in amplitude over time and within defined thresholds, following the Gaussian curve around a midpoint, called "offset". Switching the offset from zero towards positive current strength, e.g.1 mA inhibits negative polarisation during the oscillations and provides a unidirectional current flow. It is well-known that when the neurons are stimulated under a constant electrical field, the neuronal membranes adapt themselves and return to their original resting state (i.e., homeostasis of system or the homeostatic phenomena of ion neuron channels). Given the nature of constantly changing electrical field of tRNS, a potential advantage of this type of NIBS is that it might not result in homeostasis of the neural system, the mechanism thought to account for the limit to additional increases in cortical excitability with prolonged constant electrical stimulation. The pilot study in humans reported that tRNS does not work in a polarity dependent way and can increase cortical excitability under both electrodes placed on the scalp. Specifically, tRNS over the motor area positively modulates cortical excitability and improves motor learning, possibly through the mechanism of long-term potentiation (LTP). Given the particular wave shape of tRNS, it might induce temporal summation of small depolarizing currents, which could interact with the activity of the engaged neurons and therefore improve performance in perceptual learning. Therefore, tRNS of neurons provides the driving force for a synaptic potentiation-like phenomenon. The effect was more pronounced with high frequency (hf)-tRNS, which was possibly related to the range of frequency applied (100-640 Hz). Since the time constant of the neuronal cell body and dendrites has been known between 1-10 ms, stimulation at the frequency range between 100-1000 Hz may be appropriate for exerting a meaningful effect on neuronal communication. In addition, a prolonged opening of the voltage-gated sodium channels is also a possible underlying neuronal correlate for hf-tRNS to elicit more cortical excitability shifts and more pronounced plasticity changes. Another proposed mechanism through which tRNS exerts behavioral effects is the stochastic resonance phenomenon. tRNS represents a stimulation that gives rise to nonfinalized random activity in the system i.e., noise. In a linear system, noise generally reduces behavioral performance, but non-linear systems (e.g., the brain) may apply noise to improve performance via stochastic resonance. That is, neurons become sensitive to a specific range of weak inputs in the presence of an optimal level of neuronal noise, and the behavioral performance is therefore facilitated. To the investigator's knowledge, the treatment of schizophrenia with tRNS has only been reported in case studies as an add-on treatment for negative symptoms in a medicated patient or as a monotherapy in alleviating delusions and enhancing insight of the illness in a drug-free patient.

The study aimed to investigate the effects of add-on high-definition high-frequency transcranial random noise stimulation over bilateral prefrontal cortex on negative symptoms and other psychopathological symptoms, clinical outcomes (insight levels, psychosocial functioning, quality of life, beliefs about medication adherence, severity of extrapyramidal symptoms, neurocognitive function), autonomic functioning ,and brain oscillatory activity in schizophrenia patients.

Study design: randomized double-blind, sham-controlled study design.

Participants: 36 patients having a diagnosis of schizophrenia or schizoaffective were randomly allocated to receive 20 minutes of active 2-mA HD-hf-tRNS or sham stimulation twice a day on 5 consecutive weekdays. These participants were assessed at baseline, after intervention, one-week and one-month follow-ups.

Active or sham stimulation: tRNS was delivered by a battery-operated device (Eldith DC stimulator Plus, neuroConn, Ilmenau, Germany) via 5 carbon rubber electrodes (1 cm radius, high-definition 4 × 1 rings configuration with a gel layer of 2.0 mm), with 2 mA amplitude, offset at 1 mA, frequency 100-640 Hz, for 20 min with 15 s ramp-in/ramp-out. The combined impedance of all electrodes was kept below 15 kΩ, as measured by NeuroConn DC stimulator Plus device, using electrolyte gel. The anode was placed over International 10-10 electrode position AF3 (a point midway between F3 and Fp1), with cathodes (reference electrodes) at AF4, F2, F6 and FC4. The sessions were conducted twice a day on 5 consecutive working days. In the sham group, current was applied for 30 s after upward ramping and then terminated. Immediately after the first stimulation session, all participants were asked to answer the question of whether they received active or sham treatment.

Others: see Arms and Interventions, Eligibility Criteria or Outcome Measures.

ELIGIBILITY:
Inclusion Criteria:

1. Eligible participants aged 20-65 with DSM-V-defined schizophrenia or schizoaffective disorder.
2. Duration of illness ≧ 1 year.
3. Being on an adequate therapeutic dose of antipsychotics for at least 8 weeks prior to enrolment.
4. Positive and Negative Syndrome Scale (PANSS scale) total score < 120 (at both screening and baseline).
5. Agreement to participate in the study and provide the written informed consent.

Exclusion Criteria:

1. Having current psychiatric comorbidity or active substance use disorder, in exception to caffeine and/or tobacco.
2. Having a history of seizures.
3. Having contraindications for transcranial electrical stimulation or transcranial magnetic stimulation, e.g., implanted brain medical devices or metal in the head.
4. Having a history of intracranial neoplasms or surgery, or a history of severe head injuries or cerebrovascular diseases.
5. Pregnancy or breastfeeding at enrollment.

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2018-10-24 (Actual); Primary Completion 2019-05-17 (Actual); Study Completion 2019-05-17 (Actual)

PRIMARY OUTCOMES:
Changes from baseline negative dimension score of Positive and Negative Syndrome Scale (PANSS) at the timepoint immediately after HD hf-tRNS, at one-week and one-month follow-ups. | One month
  A clinician-administered rating scale to measure the severity of psychopathological symptoms of the patients with schizophrenia spectrum disorder. The patient is rated from 1 to 7 on 30 different symptom items. All items scores are summed up to yield a total PANSS score, which ranges from 30 to 210. A higher score indicates greater psychopathological symptom severity. Then, five main symptom dimension subscales of PANSS can be calculated from 26 of 30 items of PANSS: positive (5 items, score 5-35) , negative (8 items, score 8-56), grandiosity/excitement (4 items, score 4-28), disorganization (5 items, score 5-35), and depression (4 items, score 4-28).

SECONDARY OUTCOMES:
Changes from baseline scores at Personal and Social Performance scale (PSP) at the timepoint immediately after HD hf-tRNS, at one-week and one-month follow-ups. | One month
  A clinician-administered rating scale to measure the psychosocial functioning of the patients with schizophrenia spectrum disorder. The PSP scale measures psychosocial functioning within four domains: socially useful activities, personal and social relationships, self-care, and disturbing and aggressive behavior.The patient is rated from 1 to 6 on each item of the four domains. A higher score indicates greater psychosocial functioning in any of the four domains.
  The final global score is defined according to a summary instruction table. This scale provides a single, overall rating from 1 to 100, where a higher score represents better personal and social function.
Changes from baseline scores of the Global Assessment of Functioning (GAF) Scale of the DSM-IV at the timepoint immediately after HD hf-tRNS, at one-week and one-month follow-ups. | One month
  GAF is a numeric scale used by mental health clinicians and physicians to rate subjectively the social, occupational, and psychological functioning of an individual, e.g., how well one is meeting various problems-in-living. Scores range from 100 (extremely high functioning) to 1 (severely impaired). GAF serves as a valid tool of assessing global psychosocial and occupational functioning for schizophrenia patients.
Changes from baseline scores of the Clinical Global Impression (CGI) rating scales at the timepoint immediately after HD hf-tRNS, at one-week and one-month follow-ups. | One month
  Illness severity was assessed with the Clinical Global Impression (CGI) rating scales. The Clinical Global Impression
  - Severity scale (CGI-S) is a 7-point scale that requires the clinician to rate the severity of the patient's illness at the time of assessment, relative to the clinician's past experience with patients who have the same diagnosis. The patient is rated from 1 to 7 and a higher score indicates greater illness severity.
Changes from baseline scores of the self-reported version of the graphic personal and social performance scale (SRGPSP) at the timepoint immediately after HD hf-tRNS, and at one-week follow-up. | One week
  The SRG-PSP is a self-rating scale of proven validity and reliability, comprising both male and female versions of cartoon-like pictures that are derived from the narrative text of the four domains of Personal and Social Performance (PSP) scale including the sub-items of socially useful activities, personal and social relationships, self-care, and disturbing and aggressive behaviour.
Changes from baseline scores of the abbreviated version of the Scale to Assess Unawareness in Mental Disorder in schizophrenia (SUMD) at the timepoint immediately after HD hf-tRNS, at one-week and one-month follow-up. | One month.
  An expert-rating scale based on a patient interview to measure patients' clinical insight. The abbreviated version of SUMD comprises 9 items measuring current states of awareness as follows: (1) a mental disorder, (2) consequences of a mental disorder, (3) effects of drugs, (4) hallucinatory experiences, (5) delusional ideas, (6) disorganized thoughts, (7) blunted affect, (8) anhedonia, and (9) lack of sociability. Scores on each item range from 0 to 3. A score of 0 indicates 'not applicable'; 1, 'aware'; 2, 'somewhat aware/unaware' and 3, 'severely unaware.' Based on the 3 dimensions approach of the abbreviated version of SUMD, the scores on the items 1-3, 4-6 and 7-9 were averaged to obtain the dimension score of 'awareness of the disease', 'awareness of positive symptoms', and 'awareness of negative symptoms', respectively. All dimension scores were linearized on a 0-100 scale, with 0 and 100 indicating the lowest and highest level of unawareness, respectively.
Changes from baseline scores of the Taiwanese version of the Beck Cognitive Insight Scale (BCIS) at the timepoint immediately after HD hf-tRNS, and at one-week follow-up. | One week
  Cognitive insight was measured by the Taiwanese version of the Beck Cognitive Insight Scale (BCIS), a self-reported instrument comprising 15 items.The Taiwanese BCIS is composed of 2 subscales including reflective attitude (9 items) and certain attitude (6 items). We obtained a R-C (reflective attitude minus certain attitude) index of the Taiwanese BCIS, representing the measurement of cognitive insight by subtracting the score of the certain attitude subscale from that of the reflective attitude subscale. Lower R-C index scores indicate poorer cognitive insight.
Changes from baseline scores of the Taiwanese version of the Self-Appraisal of Illness Questionnaire (SAIQ) at the timepoint immediately after HD hf-tRNS, and at one-week follow-up. | One week
  The Taiwanese version of the Self-Appraisal of Illness Questionnaire (SAIQ) was used to assess attitudes toward mental illness and experience of psychiatric treatment.This self-administered tool was composed of 17 items. The patients rated the extent to which they agreed with each statement of the item by using a four-point Likert scale, ranging from 1, ''do not agree at all'', to 4, ''completely agree''. Whether the scale score is in order from least to most or from the most to least depends on the content of the item statement. The total score of SAIQ ranges from 17 to 68.
  This translated SAIQ comprises a three-factor explanation. The three factors correspond to worry (score 7-28), the need for treatment (score 5-20), and presence/outcome (score 5-20) subscales. Higher SAIQ subscale scores indicate more awareness of mental illness.
Changes from baseline scores of the self-administered WHOQOL-BREF at the timepoint immediately after HD hf-tRNS, and at one-week follow-up. | One week
  The overall quality of life (QoL) and the specific domains of QoL was measured with the self-administered World Health Organization Questionnaire on Quality of Life: Short Form-Taiwan version (WHOQOL-BREF) which was developed by the WHO in 1998 and was adapted to Taiwan's culture. The WHOQOL-BREF is of well-established validity and reliability, containing 28 five-point Likert items that assessed general (two items) and four specific domains of QoL, including 7 items in physical health, 6 in psychological, 4 in social relationships, and 9 in environmental domains. Higher scores indicate a better QoL.
Changes from baseline results of Digit span (forward and backward) at the timepoint immediately after HD hf-tRNS, and at one-week follow-up. | One week
  A test to measure the capacity of working memory of the patients.
Changes from baseline results of Finger tapping test at the timepoint immediately after HD hf-tRNS, and at one-week follow-up. | One week
  A neuropsychological test that examines motor functioning, specifically, motor speed and lateralized coordination.
Changes from baseline results of Continuous Performance (CPT, version 2.0) at the timepoint immediately after HD hf-tRNS, and at one-week follow-up. | One week
  A neuropsychological test that examines the performance of prefrontal-mediated task.
Changes from baseline results of Wisconsin Card Sorting Test (WCST) at the timepoint immediately after HD hf-tRNS, and at one-week follow-up. | One week
  A neuropsychological test of "set-shifting", i.e. the ability to display flexibility in the face of changing schedules of reinforcement.
Changes from baseline results of Tower of London test at the timepoint immediately after HD hf-tRNS, and at one-week follow-up. | One week
  A neuropsychological test for the assessment of executive functioning specifically to detect deficits in planning, which may occur due to a variety of medical and neuropsychiatric conditions.
Changes from baseline heart rate variability (HRV) at the timepoint during the first session of HD hf-tRNS, immediately after the first session of HD hf-tRNS, after the 10th session of HD hf-tRNS. | 5 days
  An index of autonomic functioning. The ECG signals were acquired, stored, pre-processed according to the recommended procedures [36] and processed by an HRV analyser (LR8Z11, Yangyin Corp., Taipei, Taiwan). The power spectrum of HRV was quantified into the standard frequency-domain measurements including variance (variance of R-R-interval values), very low-frequency power (VLF, 0.003-0.04 Hz), low-frequency power (LF, 0.04-0.15 Hz), high-frequency power (HF, 0.15-0.40 Hz), the ratio of LF/HF, normalized HF (HF%) and LF (LF%).
Changes from baseline scores of the Mini-Mental State Examination (MMSE) at the timepoint immediately after HD hf-tRNS, and at one-week follow-up. | One week
  Global cognition was assessed with the Mini-Mental State Examination (MMSE).
Changes from baseline results of Color Trails Test (CTT) at the timepoint immediately after HD hf-tRNS, and at one-week follow-up. | One week
  The CTT, a culture-neutral version of the Trail Making Test, was selected to measure sustained visual attention. The CTT consists of two parts (CTT-1 and CTT-2). The CTT-1 requires participants to connect a series of numbered circles that are randomly printed on a sheet of paper. In the CTT-2, numbered circles of 1 to 25 are shown twice (printed in pink and in yellow) randomly on a sheet of paper. Participants are asked to connect the numbers from 1 to 25 alternating between the two colors.
Changes from baseline results of Stroop Color Word Test (SCWT) at the timepoint immediately after HD hf-tRNS, and at one-week follow-up. | One week
  Stroop Color Word Test (SCWT), Chinese version; was administered to measure selective attention and cognitive flexibility. SCWT is composed of three parts, each lasting for 45 seconds.
Changes from baseline scores of Medication Adherence Rating Scale (MARS) at the timepoint immediately after HD hf-tRNS, and at one-week follow-up. | One month
  The Taiwanese version of Medication Adherence Rating Scale (MARS), translated from the original MARS, was used to assess patients' beliefs about medication adherence. The translated MARS contains 10 yes/no items. Item 1-5 formed the medication adherence subscale and item 6-10 formed the subjective response to taking medication subscale. The scores from MARS subscales were summed to yield a total MARS score ranging from 0 (poor adherence to treatment) to 10 (good adherence to treatment), indicating a broad measure of medication compliance.
Changes from baseline total scores of Extrapyramidal Symptoms Rating Scale (ESRS) at the timepoint immediately after HD hf-tRNS, at one-week and one-month follow-ups. | One month
  The Extrapyramidal Symptoms Rating Scale (ESRS) total score was used to quantitatively measure antipsychotic-induced movement disorders including Parkinsonism, akathisia, dystonia, and tardive dyskinesia. The ESRS 41 items includes 7 items of Subscale I (questionnaire), 17 items of Subscale II (Parkinsonism/Akathisia), 10 items of Part III (dystonia), and 7 items of Part IV (dyskinesia). For inter-rater reliability certification, the ESRS 41 item total score also includes the 4 CGI-S's and thus becomes ESRS 45 item total. The ESRS total score ranges from 0 to 257.
Changes from baseline values of electroencephalogram absolute power of the Delta, Theta, Alpha, Beta and Gamma frequency bands at the timepoint during and immediately after the first session of HD hf-tRNS, and after the 10th session of HD hf-tRNS. | 5 days
  In a recliner in a dimly lit, electrically shielded room, patients' resting EEGs were recorded before (baseline) and immediately after the first session of HD hf-tRNS and 3 hours after the final session of HD hf-tRNS by using the Neuro Prax® TMS/tDCS full-band DC-EEG system with 32 electrodes in the standard 10-20 International placement. EEG Ag/AgCl electrodes and HD hf-tRNS electrodes were mounted in a custom-made elastic cap for 64 electrodes. Data were collected eyes-closed and collection took ~ 10 mins and amplified in the dynamic input range of ± 140 mV at a resolution of 0.5 μV by using EEG amplifiers and stored for offline analyses. Eye or muscle artifacts were automatically detected and removed using NeuroPrax's built-in software. For the real-time recording of EEG during the first session of HD hf-tRNS, a closed-loop stimulation protocol and removal of tRNS-artefacts by using NeuroPrax's built-in algorithm were applied.

CONTACTS AND LOCATIONS:
Overall Officials: Hsin-An Chang, M.D., Principal Investigator — Tri-Service General Hospital, National Defense Medical Center
Locations (1):
- Tri-service general hospital, Taipei, Taiwan

REFERENCES:
- [Derived] Chang CC, Lin YY, Tzeng NS, Kao YC, Chang HA. Adjunct high-frequency transcranial random noise stimulation over the lateral prefrontal cortex improves negative symptoms of schizophrenia: A randomized, double-blind, sham-controlled pilot study. J Psychiatr Res. 2021 Jan;132:151-160. doi: 10.1016/j.jpsychires.2020.10.008. Epub 2020 Oct 16. PMID 33096356